CLINICAL TRIAL: NCT02764242
Title: Evaluating the Causative Insects in the Cases With Severe Insect Sting Allergy
Brief Title: The Causative Insects in Severe Insect Sting Allergy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Nualanong Visitsunthorn, Professor, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Si063/2557
Record Dates: First submitted 2016-05-04; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Insect Sting Allergy
Keywords: insect sting allergy; recombinant venom allergen
MeSH Terms: conditions — Venom Hypersensitivity | interventions — Patch Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- insect sting allergy (Other): Skin prick tests to local and imported insect sting allergen with different concentration are performed.
  sIgE Measurement (to insect and the recombinant venom)
  Interventions: Other: Skin prick test; Other: sIgE measurement

INTERVENTIONS:
Other: Skin prick test — Skin prick tests to local and imported insect sting allergen with different concentration are performed.
Other: sIgE measurement — sIgE levels to stinging insect allergen and their recombinant venom allergen are measured

SUMMARY:
Study the causative insect by skin prick test and sIgE to wasp, bee and fire ants are important but false positive by crossreactivity can occur. sIgE to recombinant venom allergen is proposed to help in finding the causative insect.

DETAILED DESCRIPTION:
Insect sting allergy from insects in Hymenoptera is not uncommon. The reaction maybe very severe and life threatening. To find the cause of insect sting allergy is important in prevention and specific treatment such as immunotherapy. The skin prick test and sIgE of these insects may have cross reactions so it is difficult to be interpreted.

The usage of sIgE recombinant venom allergen can benefit in separate cross reaction and dual allergy reaction.

ELIGIBILITY:
Inclusion Criteria:

* Cases with severe insect sting allergy reactions

Exclusion Criteria:

* Without other severe systemic diseases
* Not pregnant or lactation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-02; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Mean wheal diameters of skin prick test of local and imported insect allergens | 12 months
  Compare Mean wheal diameters of skin prick test of local and imported insect allergens at different concentrations

SECONDARY OUTCOMES:
specific IgE level to stinging insect allergen and recombinant venom allergens | 12 months
  compare skin prick test result and levels of specific IgE level to stinging insect allergen and recombinant venom allergens

IPD SHARING:
Plan to Share IPD: No